CLINICAL TRIAL: NCT00288535
Title: Prospective, Randomized, Single-Center Evaluation of the Cypher™ Sirolimus Eluting Coronary Stent System in the Treatment of Bifurcated Coronary Lesions
Brief Title: Treatment of Bifurcated Coronary Lesions With Cypher™-Stent
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Heart Center Freiburg - Bad Krozingen (Other)
Collaborators: Cordis, Johnson&Johnson company (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HZ-BK-2005-1
Record Dates: First submitted 2006-02-07; First posted 2006-02-08 (Estimated); Last update posted 2007-09-18 (Estimated); Status verified 2005-03

CONDITIONS: Coronary Artery Disease
Keywords: coronary bifurcation ; PCI; modified T-Stenting; sirolimus stent
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Procedure: PCI of bifurcated coronary lesions using sirolimus coated stents in modified T-Stenting -Technique

SUMMARY:
This study is a prospective, randomized, single-center evaluation of the Cypher™ Sirolimus eluting coronary stent system in the treatment of de novo bifurcated coronary lesions comparing provisional modified T stenting with systematic modified T-stenting.

DETAILED DESCRIPTION:
Bifurcations involving a significant side branch (SB diameter ≥ 2.25 mm) occur in approximately 15-20% of all coronary lesions considered for percutaneous intervention. If a side branch (SB) subtends significant myocardium, failure to preserve SB vessel patency can lead to complications such as myocardial infarction or persistent chest pain despite full patency of the main branch.

Bifurcation lesions are inherently complex and interventional treatment remains a challenging problem for physicians.

The optimal technique for stenting bifurcated lesions is still unknown. Several dual vessel stenting techniques have been described in the literature, such as "T", "V", "Y", "Culotte" and "Crush" procedures. However, most studies of bifurcation stenting have found that optimal long-term results are obtained by stenting the main vessel and then performing plain balloon angioplasty of the side branch ("kissing balloon"-technique). Nevertheless, occlusion or reduced flow of the SB are frequent after stenting of the MB. Therefore, the SB is stented in approximately 50% of procedures even if PTCA alone was intended.

Hypothesis:

Compared with plain dilatation of side branch, the placement of Cypher-Stent in side branch using modified T-stenting technique will reduce "in-segment percent diameter stenosis" of the side branch at 9 months post procedure as measured by quantitative coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* 1. The target vessel must meet the following criteria:

  1. Bifurcated lesion Type 1, 2, 3 or 4 of a native coronary artery with a reference vessel diameter of 2.5 mm to 4.0 mm in the main branch and of ≥ 2.25 mm in the side branch.
  2. The target lesion (main branch and / or side branch) must be at least 50% diameter stenosis.
  3. The target lesion has not been previously treated with any interventional procedure.
  4. The target vessel (main branch and side branch) must be feasible for stent implantation (successful passage with the guide wire; successful predilatation with an appropriately sized balloon; no heavy calcification; no diffuse distal disease that might impede run off).

     2. Patient has stable or unstable angina pectoris (CCS classification I or greater) or a positive stress test for ischemia.

     3. Patient must be ≥ 18 years of age. 4. Female subjects of childbearing potential must have a negative pregnancy test within 7 days before the procedure.

     5. Patient has no other treatment planned within 30 days of the procedure. 6. Patient has been informed of the nature of the study and agrees to its provisions and has written informed consent as approved by the Ethics Committee.

     7. Patient willing to comply with required post-procedure follow-up.

     Exclusion Criteria:
* 1. Patient has had an acute myocardial infarction (> 3x normal CK with presence of CKMB) within 72 hours preceding the index procedure and CK has not returned to normal limits at the time of the procedure.

  2. Patient will have a known hypersensitivity or contraindication to aspirin, heparin, clopidogrel, stainless steel, sirolimus, or contrast sensitivity that cannot be adequately pre-medicated.

  3. Patient has a platelet count of <100,000 cells/mm³ or >700,000 cells/mm³, a WBC of <3,000 cells/mm³, or documented or suspected liver disease.

  4. Patient has a history of bleeding diathesis or coagulopathy. 5. Patient has suffered a CVA or TIA within the past six months. 6. Active peptic ulcer or upper GI bleeding within the prior 6 months. 7. Patient has a co-morbidity (i.e. cancer or congestive heart failure) that may cause the patient to be non-compliant with the protocol, or is associated with limited life- expectancy (less than 2 years).

  8. Patient must be excluded from the study if any of these angiographic criteria are met:
  1. The target vessel contains intraluminal thrombus.
  2. The target lesion is located in the left main coronary artery.
  3. The target lesion or vessel shows angiographic evidence of severe calcification.
  4. The patient has undergone previous PCI to the target vessel within 6 months.
  5. Pre treatment of the lesion is done with a technique other than balloon angioplasty (e.g. rotablation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2005-03; Study Completion 2007-02

PRIMARY OUTCOMES:
In-segment percent diameter stenosis of the side branch at 9 months post procedure as measured by quantitative coronary angiography.

SECONDARY OUTCOMES:
Freedom from Major Adverse Cardiac Events (MACE)at 30 days, 6 and 12 months
Angiographic binary restenosis (≥ 50% diameter stenosis) in the main and side branch at 9 months post procedure.
Target Lesion Revascularization (TLR) at 12 months post procedure.
Device success during PCI
Post-procedure thrombotic stent occlusion at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Miroslaw FERENC, Dr., Principal Investigator — Haert Center Bad Krozingen; Germany; Franz-Josef Neumann, Prof. Dr., Study Director — Heart Center Bad Krozingen, Germany
Locations (1):
- Herz-Zentrum Bad Krozingen, Bad Krozingen, Suedring 15, Germany

REFERENCES:
- [Background] Colombo A, Moses JW, Morice MC, Ludwig J, Holmes DR Jr, Spanos V, Louvard Y, Desmedt B, Di Mario C, Leon MB. Randomized study to evaluate sirolimus-eluting stents implanted at coronary bifurcation lesions. Circulation. 2004 Mar 16;109(10):1244-9. doi: 10.1161/01.CIR.0000118474.71662.E3. Epub 2004 Feb 23. PMID 14981005
- [Background] Lefevre T, Louvard Y, Morice MC, Dumas P, Loubeyre C, Benslimane A, Premchand RK, Guillard N, Piechaud JF. Stenting of bifurcation lesions: classification, treatments, and results. Catheter Cardiovasc Interv. 2000 Mar;49(3):274-83. doi: 10.1002/(sici)1522-726x(200003)49:33.0.co;2-n. PMID 10700058
- [Background] Al Suwaidi J, Yeh W, Cohen HA, Detre KM, Williams DO, Holmes DR Jr. Immediate and one-year outcome in patients with coronary bifurcation lesions in the modern era (NHLBI dynamic registry). Am J Cardiol. 2001 May 15;87(10):1139-44. doi: 10.1016/s0002-9149(01)01482-5. PMID 11356386
- [Background] Holmes DR, Leon MB, Moses JW et al. One-year follow-up of the SIRIUS study : a randomized study with the sirolimus-eluting Bx Velocity in the treatment of patients with denovo native coronary artery lesions. J Am Coll Cardiol 2003;41:32A
- [Background] Yamashita T, Nishida T, Adamian MG, Briguori C, Vaghetti M, Corvaja N, Albiero R, Finci L, Di Mario C, Tobis JM, Colombo A. Bifurcation lesions: two stents versus one stent--immediate and follow-up results. J Am Coll Cardiol. 2000 Apr;35(5):1145-51. doi: 10.1016/s0735-1097(00)00534-9. PMID 10758954
- [Derived] Ferenc M, Ayoub M, Buttner HJ, Gick M, Comberg T, Rothe J, Valina CM, Hochholzer W, Neumann FJ. Long-term outcomes of routine versus provisional T-stenting for de novo coronary bifurcation lesions: five-year results of the Bifurcations Bad Krozingen I study. EuroIntervention. 2015 Dec;11(8):856-9. doi: 10.4244/EIJV11I8A175. PMID 26696453
- [Derived] Ferenc M, Gick M, Kienzle RP, Bestehorn HP, Werner KD, Comberg T, Kuebler P, Buttner HJ, Neumann FJ. Randomized trial on routine vs. provisional T-stenting in the treatment of de novo coronary bifurcation lesions. Eur Heart J. 2008 Dec;29(23):2859-67. doi: 10.1093/eurheartj/ehn455. Epub 2008 Oct 9. PMID 18845665